CLINICAL TRIAL: NCT05394389
Title: The Complementary Contributions of Sensory Stimulation and Social Support During Snoezelen Room Therapy on the General Physical and Emotional Health of the Elderly Population: Optimization of the Nursing Home Resources.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pavel Goldstein (Other)
Responsible Party: Sponsor-Investigator, Pavel Goldstein, Head of Integrative Pain Laboratory, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Upshaifa
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Loneliness; Aging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sensory-stimulating therapy (Active Comparator)
  Interventions: Other: sensory stimulating therapy
- social interaction (Active Comparator)
  Interventions: Other: social support
- combined sensory-stimulating therapy and social interaction. (Experimental)
  Interventions: Other: sensory stimulating therapy; Other: social support

INTERVENTIONS:
Other: sensory stimulating therapy — therapy session in the snoozlen room accompanied by social support.
  Other Names: integrative approach sensory stimulating therapy and social support
  Arms: combined sensory-stimulating therapy and social interaction.; sensory-stimulating therapy
Other: social support — ten minutes of conversing.
  Arms: combined sensory-stimulating therapy and social interaction.; social interaction

SUMMARY:
Over time, lifespan is extending, the population is aging, and accordingly there is a great demand for hospital beds in nursing homes, increasing attention to this population and the services they receive. Mostly, elderly population living in nursing homes suffers from dementia, Alzheimer, depression, agitation, and other diseases that require multidisciplinary treatment.

In addition to the medical and pharmacological treatments that patients receive to maintain functional medical status, there is a great need for non-pharmacological treatments, that may improve quality of life, mental well-being, and life satisfaction.

There are several treatment approaches of multisensory stimulation environment (MSSE). MSSE in the Snoezelen room therapy recognized as benefiting the patients' physical, mental, and emotional health status. In addition, there is great importance of intervention by social interaction, support, and encouragement.

However, the effect of combined intervention of MSSE in Snoezelen room therapy and social support, has not yet been sufficiently studied in elderly patients in nursing homes. These two interventions - together - are supposed to have an increased effect on physical and mental wellbeing of elderly.

ELIGIBILITY:
Inclusion Criteria:

* Patients living in the Ahuzat Moriah nursing home\ geriatric nursing hospital in Shefar'am.

Exclusion Criteria:

* Patients with epilepsy and aggressive patients. *We do not limit the participation of patients whose cognitive level is very low.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
pain, patient- reported outcome, measured by a ruler from zero to 10, on the Likert scale | four weeks
  An interval variable measured by a ruler from zero to 10, on the Likert scale, and with the help of illustrations of faces, the farther away from zero, the higher the intensity of pain.
grip strength | eighteen minutes
  A continuous quantitative variable presented in numerical values of isometric grip force from 0 to 90 kg and will be measured by Jamar hydraulic dynamometer. The hand grip strength will be measured in a hydraulic dynamometer borrowed from the university. The assessment does not involve any potential damage, a two-minute test in which the subject is required to press a device to measure grip strength.
life satisfaction, patient-reported outcome. | four weeks
  using the SWLS questionnaire before the first session and after the fourth(last) session as an estimation tool .Interval variable, showing scores ranging from 5-35, on the Likert scale, the higher the score it indicates more life satisfaction.
general anxiety disorder, patient- reported outcome | four weeks
  using the GAD questionnaire before the first session and after the fourth(last) session as an estimation tool.GAD- is an interval variable, which will be measured using the sum of the reports on the 7 statements on the Likert scale from 0 to 3, the higher the score on this questionnaire, the higher the level of anxiety among the patient. The total score range is from 0-21.
blood pressure | eighteen minutes
  Continuous quantitative variable, will be measured by a blood pressure monitor "Welch Allyn" measuring instrument\ device and quantitatively represented, this result variable will examine the quantitative change in systolic and diastolic blood pressure.

SECONDARY OUTCOMES:
pulse(heart rate index) | eighteen minutes
  Continuous quantitative variable, will be measured by "Welch Allyn" measuring instrument\ device.
oxygen saturation | eighteen minutes
  Continuous quantitative variable, will be measured by "Welch Allyn" measuring instrument\ device. and presents the degree of oxygen concentration in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahuzat Moriah Shfraam, Haifa, North, Israel

REFERENCES:
- [Derived] Khatib S, Palgi Y, Ashar YK, Polyvyannaya N, Goldstein P. The Combined Effect of Multisensory Stimulation and Therapist Support on Physical and Mental Health of Older Adults Living in Nursing Homes: Pilot Randomized Controlled Trial. J Med Internet Res. 2025 Jan 14;27:e55042. doi: 10.2196/55042. PMID 39808474